CLINICAL TRIAL: NCT00860938
Title: Predictor for an Additional Benefit of Inhaled Corticosteroid in Patients Treated With Tiotropium for Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Predictor for an Additional Benefit of Inhaled Corticosteroid in Patients Treated With Tiotropium for COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cantonal Hosptal, Baselland (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jörg Leuppi, Prof. Dr., Cantonal Hosptal, Baselland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EKBB 148/06
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: COPD
Keywords: Inhaled corticosteroids; COPD; mannitol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Budesonide (Active Comparator)
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator)
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — After 4 weeks of inhalative therapy with tiotropium (all patients), patient get randomized to receive either inhalative budesonide (1600ug per day or placebo
  Other Names: Miflonide

SUMMARY:
Study purpose is to evaluate if subjects with chronic obstructive pulmonary disease (COPD) are more likely to be responsive to additional inhaled corticosteroids if they have a positive response to hyperosmolar challenge with mannitol than if their response is negative.

DETAILED DESCRIPTION:
In patients with chronic obstructive pulmonary disease (COPD), the treatment with inhaled corticosteroids (ICS) is controversial. Preliminary results of our recent pilot study in 30 COPD patients showed for the first time, that ICS response mey be predicted by a bronchoprovocation challenge test with mannitol. However, this finding needs to be proven in a placebo-controlled trial. For this cohort study, 100 corticosteroid-naive, non reversible (FEV1) patients with COPD will be recruited. Spirometry before and after bronchodilation will be measured at study entry and at four weeks run-in (only tiotropium) and at three month of treatment with tiotropium and ICS or placebo. Quality of life (St. George Respiratory Quality of Life Questionnaire) and exacerbation rate of COPD will be assessed. Measurement of exhaled nitric oxide and mannitol challenge will be performed at study entry and at 1 and 4 month. Primary endpoint will be improvement in FEV1 in each group (positive and negative mannitol challenge) after 3 months follow up. Secondary endpoints will be the difference in dose-response-curve in the mannitol challenge, exacerbation rate and change in quality of life after three month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* FEV1/FVC < 70%
* FEV1 % predicted > 60%

Exclusion Criteria:

* Other major disease
* Asthma
* Currently taking inhaled corticosteroids
* oral corticosteroids in the last 3 month
* significant cardiovascular disease
* pregnancy/breast feeding
* current use of salmeterol or other long acting bronchodilator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-04; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jörg D Leuppi, MD PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Scherr A, Schafroth Torok S, Jochmann A, Miedinger D, Maier S, Taegtmeyer AB, Chhajed PN, Tamm M, Leuppi JD. Response to add-on inhaled corticosteroids in COPD based on airway hyperresponsiveness to mannitol. Chest. 2012 Oct;142(4):919-926. doi: 10.1378/chest.11-2535. PMID 22459771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: out patient clinic
Pre-assignment Details: run-in
Period: Overall Study
Arm/Group | Budesonide | Placebo
Started | 45 | 45
Completed | 31 | 37
Not Completed | 14 | 8

BASELINE CHARACTERISTICS:
Population: We recruited 90 participants as per protocol. However, inclusion had to be stopped for organisational reasons when 31 patients in the budesonide and 37 on the Placebo group were recruited.
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide | Placebo | Total
Number analyzed (Participants) | 31 | 37 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 18 | 23 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (16) | 62 (22) | 61.5 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 31
  Male | 19 | 18 | 37
Region of Enrollment [Number; unit: participants]
  Switzerland | 31 | 37 | 68
FEV1/FVC [Mean (Standard Deviation); unit: %] | 63 (10) | 64 (10) | 64 (10)

OUTCOME MEASURES:

1. Primary Outcome: Change in Lung Function (FEV1)
Time Frame: 12 weeks
Population: per protocol
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 31 | 37
litres | 0.05 (0.01) | -0.05 (0.01)

2. Secondary Outcome: The Proportion Who Complete Follow-up Without Developing an Exacerbation
Time Frame: 12 weeks
Measure: Number; unit: number of participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 31 | 37
number of participants | 31 | 37

3. Secondary Outcome: Change in Quality of Life
Description: St. George Respiratory Questionnaire (SGRQ). Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.
  Scores are calculated for three domains: Part I (Symptoms): several scales; Part II (Activity and Impacts): dichotomous (true/false) except last question (4-point Likert scale) Scores range from 0 to 100, with higher scores indicating more limitations. Unit of Measure = Units on a scale A minimum change in score of 4 units was established as clinically relevant after patient and clinician testing.
  Based on empirical data and interviews with patients, a mean change score of 4 units is associated with slightly efficacious treatment, 8 units for moderately efficacious change and 12 units for very efficacious treatment. The higher the change in units, the better the treatment.
Time Frame: 12 weeks, baseline to 3 months follow-up
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 31 | 37
units | 5.1 (5.8) | 1.8 (0.3)

4. Secondary Outcome: Change in logRDR Mannitol
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: %/mg
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 31 | 37
%/mg | 0.12 (0.1) | -0.09 (0.01)

ADVERSE EVENTS:
Arm/Group | Budesonide | Placebo
Serious Adverse Events (participants affected / at risk) | 1/31 | 2/37
Other Adverse Events (participants affected / at risk) | 2/31 | 2/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide (N=31) | Placebo (N=37)
Urosepsis (Renal and urinary disorders) | 1 | 2
unstable angina pectoris (Cardiac disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide (N=31) | Placebo (N=37)
Acute exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
The dropout rate of 24% was relatively high. A further limitation of the study might be the lack of data for sputum eosinophilia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes